CLINICAL TRIAL: NCT07346131
Title: ELUDYN: Assessment of Intra-individual Variability of Vascular Dynamics of Gadopiclenol Injection Parameters in Contrast-enhanced MRI
Acronym: ELUDYN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2025-01760
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Contrast Agent; Medical Imaging Data; MRI Image Enhancement
MeSH Terms: interventions — Contrast Media; Gadolinium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Injection protocol 1: gadopiclenol 2 mL/s (Experimental)
  Interventions: Drug: contrast agent, Gadolinium
- Injection protocol 2: gadopiclenol 1 mL/s (Experimental)
  Interventions: Drug: contrast agent, Gadolinium
- Injection protocol 3: gadopiclenol 0.5 mL/s (Experimental)
  Interventions: Drug: contrast agent, Gadolinium
- Injection protocol 4: gadopiclenol half dose (Experimental)
  Interventions: Drug: contrast agent, Gadolinium
- Injection protocol 5: gadoteric acid 1 mL/s (Active Comparator)
  Interventions: Drug: contrast agent, Gadolinium

INTERVENTIONS:
Drug: contrast agent, Gadolinium — Each participant undergoes five abdominal MRI exams with distinct injection protocols in a random order with at least a 2-week interval between each exams.

SUMMARY:
This study aims to understand how the volumes and speeds of intravenous injection of a recent type of contrast agent can be optimized in order to improve the information provided by medical images. To do this, five MRI scans lasting approximately 30 minutes will be performed on 10 healthy volunteers over a period of approximately 10 months. The images will then be analyzed by three radiologists who will view the images in different orders, without knowing which injection parameters were used. They will decide, based on their impressions but also on precise measurements in the images, which parameters produce the best images.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 and ≤ 40 years of age at time of Informed Consent
* Informed Consent as documented by signature
* No known chronic conditions (defined by ICD-10 codes)
* Non-smoking
* French speaking

Exclusion Criteria:

* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Contraindications to the class of drug (gadopiclenol and gadoteric acid) under study, e.g. known hypersensitivity or allergy
* Claustrophobia and contraindication for MRI according to institutional practices
* Prior MRI examination with contrast agent and washout period of ≤ 2 weeks
* Prior liver, spleen, pancreatic or bowel surgery
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational medicinal product within the 30 days preceding and during the present study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative evaluation of MRI images | June 2027
  The qualitative evaluation of the MRI images, as assessed by the median composite score of three five-items Likert scales (0 = non-diagnostic or unacceptable; 1 = poor; 2 = fair; 3 = good; 4 = excellent) across the rating of three experienced radiologists. The three Likert scales concern i) the border delineation of the vessel measured using slopes perpendicular to the vessel walls, ii) the internal homogeneity in the vessel, and iii) the visual degree of contrast enhancement. The composite score thus ranges from 0 to 12 for each reader and then the middle score (i.e., the median) between all three readers is taken for increased reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- HFR Hôpital fribourgeois, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No